CLINICAL TRIAL: NCT03249051
Title: Optimization of Nutritional Therapy by Variation of Methods to Determine Energy Needs in Mechanically Ventilated, Critically Ill Patients.
Brief Title: Optimization of Nutritional Therapy in Mechanically Ventilated, Critically Ill Patients.
Acronym: ONCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Indirect Calorimetry in ICU
Record Dates: First submitted 2017-06-25; First posted 2017-08-15 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-08

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness | interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Calorimetry (Experimental): The energy need is being determined by using indirect calorimetry and if necessary, optimized by parenteral, enteral and additive parenteral nutrition.
  Interventions: Other: Indirect Calorimetry
- Standard Care (No Intervention): This group receives nutrition supply according to the hospital routine ("standard care")

INTERVENTIONS:
Other: Indirect Calorimetry — Energy need is being determined using indirect Calorimetry
  Arms: Indirect Calorimetry

SUMMARY:
The aim of this study is to investigate whether an individualized determination of energy requirements using indirect calorimetry instead of a formula-based approach leads to an optimized nutritional support and as a consequence to an optimized nutritional status of the critically ill, mechanically ventilated patients measured by the phase angle.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* mechanical ventilation
* an hospital stay of at least three days at the intensive care unit of the University Hospital of Tübingen
* possibility to perform indirect calorimetry measurements (FiO2 ≤70, PCO2 ≤ 0,5)
* possibility to perform Bioelectrical Impedance Analysis (BIA)
* underlying indication for enteral or/and parenteral nutritional support
* written informed consent from the patient or a legal authorized person

Exclusion Criteria:

* cardiac pacemaker

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Phase angle (PhA) | PhA was measured between one and 90 days (during ICU stay)
  The primary endpoint is the change of the phase angle during the stay in the intensive care unit (ICU). A mean difference of 5% is considered as relevant.

SECONDARY OUTCOMES:
Nitrogen Balance | Nitrogen Balance was measured between one and 90 days (during ICU stay)
  Difference between intervention and control group between hospital admission and discharge.
Extracellular to body cell mass ratio (ECM/BCM - Ratio) | ECM/BCM-Ratio was measured between one and 90 days (during ICU stay)
  Difference between intervention and control group between hospital admission and discharge.
Length of hospital stay in days | Length of hospital stay was measured between one and 180 days
  Difference between intervention and control group between hospital admission and discharge.
Length of stay in intensive care unit (ICU) in days | Length of ICU stay was measured between one and 90 days
  Difference between intervention and control group between hospital admission and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, Principal Investigator — University of Hohenheim, 70599 Stuttgart, Germany
Locations (1):
- University of Hohenheim, Stuttgart, Germany